CLINICAL TRIAL: NCT06134323
Title: Efficacy and Mechanism of Transcutaneous Vagus Nerve Stimulation in the Treatment of Generalized Anxiety Disorder
Brief Title: Transcutaneous Vagus Nerve Stimulation for Generalized Anxiety Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20232271-F-1
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: medication-combined transcutaneous vagus nerve stimulation group or the medication-combined sham stimulation group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- medication-combined transcutaneous vagus nerve stimulation (Experimental): Participants will receive anti-anxiety medication and transcutaneous vagus nerve stimulation
  Interventions: Device: medication-combined transcutaneous vagus nerve stimulation
- medication-combined sham stimulation group (Placebo Comparator): Participants will receive anti-anxiety medication and sham stimulation
  Interventions: Device: medication-combined sham stimulation

INTERVENTIONS:
Device: medication-combined transcutaneous vagus nerve stimulation — Two electrodes will be applied 2 cm below the left carotid sinus for active stimulation
  Arms: medication-combined transcutaneous vagus nerve stimulation
Device: medication-combined sham stimulation — Two electrodes will be applied 2 cm below the left carotid sinus for sham stimulation
  Arms: medication-combined sham stimulation group

SUMMARY:
This is a randomized, double-blind, parallel-controlled study of patients with generalized anxiety disorder, who will be randomly assigned to either drug-combined transcutaneous vagus nerve stimulation (tVNS) group or drug-combined sham-stimulation group for a period of 4 weeks of treatment.Scale assessments will be performed at baseline, week 1, week 2, week 3, and week 4 of treatment, and brain function monitoring as well as laboratory tests will be performed at baseline and at the end of treatment, respectively.The aim of this study is to investigate the efficacy of medication combined with tVNS and the possible mechanisms of tVNS in the treatment of anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-5 diagnostic criteria for Generalized Anxiety Disorder;
* Having a first episode of Generalized Anxiety Disorder or not having used an anxiolytic, antidepressant, antipsychotic, or anticonvulsant medication in the last 1 month.
* Having a Hamilton Anxiety Scale (HAMA) score of more than 14 and a Hamilton Depression Scale (HAMD-17) score of less than 17.

Exclusion Criteria:

* Having organic brain lesions (e.g., cerebral hemorrhage, massive cerebral infarction, encephalitis, epilepsy); cardiac QTc interval > 450ms;
* Current or previous diagnosis of other major diseases (e.g., coronary heart disease, pulmonary heart disease, etc.)
* Currently or previously diagnosed with a mental disorder other than anxiety disorder (except for insomnia disorder);
* Those who are participating or have participated in vagus nerve stimulation therapy; those who are participating in transcranial magnetic stimulation or transcranial direct current therapy;
* Pregnant, breastfeeding, or planning to become pregnant during the trial;
* Refusing to sign the informed consent form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the Hamilton Anxiety Scale at Baseline and Week 2 of Treatment | Baseline and Week 2 of the treatment
  The Hamilton Anxiety Scale is a physician evaluation scale commonly used in clinical practice to assess the level of anxiety in patients. Changes in its scores accurately reflect changes in anxiety symptoms. In this study, changes in scores at baseline and the second week of treatment will be used as the primary outcome measure.

SECONDARY OUTCOMES:
Changes in the Hamilton Anxiety Scale at Baseline and Week 4 of Treatment | Baseline and Week 4 of the treatment
  The Hamilton Anxiety Scale is a physician evaluation scale commonly used in clinical practice to assess the level of anxiety in patients. Changes in its scores accurately reflect changes in anxiety symptoms.Higher scores mean that the patient's anxiety is more severe.
Changes in the Hamilton Depression Scale at Baseline and Week 2 of Treatment | Baseline and Week 2 of the treatment
  The Hamilton Depression Scale is a physician evaluation scale commonly used in clinical practice to assess the level of depression in patients. Changes in its scores accurately reflect changes in depressive symptoms.Higher scores mean that the patient is more severely depressed.
Changes in the Hamilton Depression Scale at Baseline and Week 4 of Treatment | Baseline and Week 4 of the treatment
  The Hamilton Depression Scale is a physician evaluation scale commonly used in clinical practice to assess the level of depression in patients. Changes in its scores accurately reflect changes in depressive symptoms.Higher scores mean that the patient is more severely depressed.
Changes in the Generalized Anxiety Scale at Baseline and Week 2 of Treatment | Baseline and Week 2 of the treatment
  The Generalized Anxiety Scale is a self-assessment scale commonly used in clinical practice to evaluate generalized anxiety symptoms. It has only 7 items and is easy to use.Higher scores mean that the patient's anxiety is more severe.
Changes in the Generalized Anxiety Scale at Baseline and Week 4 of Treatment | Baseline and Week 4 of the treatment
  The Generalized Anxiety Scale is a self-assessment scale commonly used in clinical practice to evaluate generalized anxiety symptoms. It has only 7 items and is easy to use.Higher scores mean that the patient's anxiety is more severe.
Changes in brain function indicators from baseline to end of treatment | Baseline and Week 4 of the treatment
  Functional near-infrared spectroscopy and event-related potentials will be used in this study to examine brain function in patients.Event-related potential (ERP) is a special brain evoked potential that is generated by intentionally giving a stimulus a special psychological meaning, using multiple or multiple stimuli. Functional near-infrared spectroscopy (fNIRS) can utilize the good scattering of 600-900nm near-infrared light by the main components of blood to obtain changes in oxyhemoglobin and deoxyhemoglobin during brain activity.
Incidence of adverse events in each group | Baseline and Week 4 of the treatment
  During the study period, any treatment-related adverse events will be recorded and used to evaluate the safety of the intervention.Common side effects include changes in pronunciation, hoarseness, neck pain, cough, vomiting, etc

CONTACTS AND LOCATIONS:
Overall Officials: Yihuan Yihuan, Principal Investigator — The First Affiliated Hospital of the Air Force Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Air Force Military Medical University, Xi'an, Shaanxi
  - Xi'an No.3 Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang Y, Wang Y, Wang H, Liu Z, Yu X, Yan J, Yu Y, Kou C, Xu X, Lu J, Wang Z, He S, Xu Y, He Y, Li T, Guo W, Tian H, Xu G, Xu X, Ma Y, Wang L, Wang L, Yan Y, Wang B, Xiao S, Zhou L, Li L, Tan L, Zhang T, Ma C, Li Q, Ding H, Geng H, Jia F, Shi J, Wang S, Zhang N, Du X, Du X, Wu Y. Prevalence of mental disorders in China: a cross-sectional epidemiological study. Lancet Psychiatry. 2019 Mar;6(3):211-224. doi: 10.1016/S2215-0366(18)30511-X. Epub 2019 Feb 18. PMID 30792114
- [Background] Slee A, Nazareth I, Bondaronek P, Liu Y, Cheng Z, Freemantle N. Pharmacological treatments for generalised anxiety disorder: a systematic review and network meta-analysis. Lancet. 2019 Feb 23;393(10173):768-777. doi: 10.1016/S0140-6736(18)31793-8. Epub 2019 Jan 31. PMID 30712879
- [Background] Bereza BG, Machado M, Ravindran AV, Einarson TR. Evidence-based review of clinical outcomes of guideline-recommended pharmacotherapies for generalized anxiety disorder. Can J Psychiatry. 2012 Aug;57(8):470-8. doi: 10.1177/070674371205700805. PMID 22854029
- [Background] Batelaan NM, Bosman RC, Muntingh A, Scholten WD, Huijbregts KM, van Balkom AJLM. Risk of relapse after antidepressant discontinuation in anxiety disorders, obsessive-compulsive disorder, and post-traumatic stress disorder: systematic review and meta-analysis of relapse prevention trials. BMJ. 2017 Sep 13;358:j3927. doi: 10.1136/bmj.j3927. PMID 28903922
- [Result] Bonaz B, Bazin T, Pellissier S. The Vagus Nerve at the Interface of the Microbiota-Gut-Brain Axis. Front Neurosci. 2018 Feb 7;12:49. doi: 10.3389/fnins.2018.00049. eCollection 2018. PMID 29467611
- [Result] Noble LJ, Meruva VB, Hays SA, Rennaker RL, Kilgard MP, McIntyre CK. Vagus nerve stimulation promotes generalization of conditioned fear extinction and reduces anxiety in rats. Brain Stimul. 2019 Jan-Feb;12(1):9-18. doi: 10.1016/j.brs.2018.09.013. Epub 2018 Sep 21. PMID 30287193